CLINICAL TRIAL: NCT03041623
Title: Japanese Idiopathic Interstitial Pneumonias Registry
Acronym: JIPS
Status: Active, not recruiting | Type: Observational
Sponsor: North East Japan Study Group (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: NEJ030
Record Dates: First submitted 2016-12-18; First posted 2017-02-03 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Interstitial Pneumonia
Keywords: IIPs
MeSH Terms: conditions — Idiopathic Interstitial Pneumonias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
An objective of JIPS Registry is to examine disease behavior of idiopathic interstitial pneumonias (IIPs), considering classification, background, and diagnostic methods based on American Thoracic Society (ATS)/ European Respiratory Society(ERS) /Japanese Respiratory Society (JRS)/ Latin American Thoracic Association (ALAT) guidelines for diagnosis and the ATS/ERS classification of 2002 and 2013.

DETAILED DESCRIPTION:
JIPS Registry is a multi-site, non-interventional, prospective observation study of patients with newly diagnosed IIPs in Japan. At least 600 patients will be registered for 16 months at approximately 80 sites in Japan.

Primary research question is to determine the natural history of each category of IIPs at registration, patient background and diagnosis methods will be considered. Furthermore, the present treatment patterns and disease behavior (CT and forced vital capacity (FVC) changes, as well as changes in interstitial pneumonia markers, etc.) will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 20 and 84 years
2. Patients with idiopathic pulmonary fibrosis (IPF) and other IIPs diagnosis within 6 months before registration at each facility
3. Patients from whom written informed consent has been obtained regarding participation in this study and follow-up observation

Exclusion Criteria:

1. Patients for whom the tests (such as the lung function test) conducted in this study could not be performed
2. Patients who underwent pulmonary resection
3. Patients undergoing dialysis
4. Patients with cancer treated at the time of registration or those planning to receive treatment in the future

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed IIPs within 6 months before registration
Sampling Method: Non-Probability Sample
Enrollment: 867 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Data on current practice patterns for diagnosis of IIPs | 3-4 years
  Describe the frequency of surgical lung biopsy, bronchoalveolar lavage.
Prevalence of each categorized IIPs | 3-4 years
  Investigate the prevalence of each categorized IIPs by using a recent guideline
Natural history of each categorized IIPs | 3-4 years
  Describe the natural history of each categorized IIPs, focusing on CT findings, FVC changes, medications, and causes of death.

SECONDARY OUTCOMES:
Progression-free survival by category of IIPs | 3-6 years
Hospital admission for acute exacerbations of IIPs | 3-6 years
  To evaluate incidences, therapy and prognosis of acute respiratory deterioration in patients with IIPs
Mean change of patient-reported outcome (Saint George Respiratory Questionnaire, COPD assessment test, and Dyspnoea-12) every12 months from baseline | 3-4 years
Quantitative evaluation of CT findings | 3-6 years
Validation of second multidisciplinary discussion | 3-4 years
  Multidisciplinary discussion (MDD) held by independent central reviewers will be conducted twice at the time of registration and final observation using questionnaire. Concordance rate for diagnosis and disease behavior in each case between the time of registration and final observation will be evaluated.
Validation of new guideline | 3-6 years
  If there are changes in IIPs diagnostic guidelines or severity classification during this study, these changes will be verified.
Diagnosis of IIPs in patients with IIPs at registration | At registration and 1 year after registration
  Describe the frequency of IIPs diagnosis using data at the time of registration.

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Ogura, MD, Principal Investigator — Kanagawa Cardiovascular and Respiratory Center
Locations (86):
- Japan (86):
  - Haruhi Respiratory Medical Hospital, Kiyosu, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Tosei General Hospital, Seto, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - Chiba University Hospital, Chiba, Chiba
  - National Hospital Organization Chiba-East-Hospital, Chiba, Chiba
  - Kameda Medical Center, Kamogawa, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - University of Fukui Hospital, Yoshida, Fukui
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Kyushu University Hospital., Fukuoka, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Aso Iizuka Hospital, Iizuka, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - University of Occupational and Environmental Health Japan, Kitakyushu, Hukuoka
  - National Hospital Organization Himeji Medical Center, Himeji, Hyōgo
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kobe City Medical Center West Hospital, Kobe, Hyōgo
  - Ibarakihigashi National Hospital, Naka, Ibaraki
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Prefectural Central Hospital, Morioka, Iwate
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Tokai University Hospital, Isehara, Kanagawa
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Showa University Fujigaoka Hospital, Yokohama, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Kochi medical School Hospital, Nankoku, Kochi
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Japanese Red Cross Ise Hospital, Ise, Mie-ken
  - Matsuzaka City Hospital, Matsuzaka, Mie-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai, Miyagi
  - Suwa Central Hospital, Chino, Nagano
  - Shinshu University Hospital, Matsumoto, Nagano
  - Saku Central Hospital Advanced Care Center, Saku, Nagano
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Tenri Hospital, Tenri, Nara
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - National Hospital Organization Minami-Okayama Medical Center, Okayama, Okayama-ken
  - Okinawa Chubu Hospital, Uruma, Okinawa
  - National Hospital Organization Kinki-chuo Chest Medical Center, Sakai, Osaka
  - Kinki University Hospital, Sayama, Osaka
  - Dokkyo Medical University Koshigaya Hospital, Koshigaya, Saitama
  - Japanese Red Cross Saitama Hospital, Saitama, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Shimane University Hospital, Izumo, Shimane
  - National Hospital Organization Matsue Medical Center, Matsue, Shimane
  - Hamamatsu Rosai Hospital, Hamamatsu, Shizuoka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Seirei Mikatahara General Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University, Shimotsuke, Tochigi
  - Dokkyo Medical University Hospital, Tochigi, Tochigi
  - Tokushima University Hospital, Tokushima, Tokushima
  - National Hospital Organization Tokyo National Hospital, Kiyose, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Toranomon Hospital, Tokyo, Tokyo
  - The Jikei University Hospital, Tokyo, Tokyo
  - Juntendo University Hospital, Tokyo, Tokyo
  - Tokyo Medical and Dental University, Tokyo, Tokyo
  - Nippon Medical School Hospital, Tokyo, Tokyo
  - Tokyo University Hospital, Tokyo, Tokyo
  - NTT Medical Center Tokyo, Tokyo, Tokyo
  - Toho University Omori Medical Center, Tokyo, Tokyo
  - Japanese Red Cross Medical Center, Tokyo, Tokyo
  - JR Tokyo General Hospital, Tokyo, Tokyo
  - National Hospital Organization Tokyo Medical Center, Tokyo, Tokyo
  - National Center for Global Health and Medicine, Tokyo, Tokyo
  - Teikyo University Hospital, Tokyo, Tokyo
  - Nihon University Itabashi Hospital, Tokyo, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Toyama University Hospital, Toyama, Toyama
  - Yamagata City Hospital Saiseikan, Yamagata, Yamagata
  - National Hospital Organization Yamaguchi-Ube Medical Center, Ube, Yamaguchi

REFERENCES:
- [Derived] Okuda R, Ogura T, Hisata S, Baba T, Kondoh Y, Suda T, Johkoh T, Iwasawa T, Tomioka H, Bando M, Azuma A, Inoue Y, Ishikawa N, Arai N, Takihara T, Hamaguchi M, Arai T, Nakamura Y, Miyamoto A, Tomii K, Miyazaki Y, Chiba H, Ishii H, Hamada N, Terasaki Y, Fukuoka J, Sakai F, Egashira R, Fujimoto K, Sumikawa H, Suzuki T, Sakamoto S, Nishioka Y, Hattori N, Hashimoto N, Morita S, Ichihara N, Miyata H, Hagiwara K, Kobayashi K, Nukiwa T; JIPS registry collaborators. Prognostic prediction for newly diagnosed patients with idiopathic interstitial pneumonia: JIPS Registry (NEJ030). Respir Investig. 2025 May;63(3):365-372. doi: 10.1016/j.resinv.2025.02.009. Epub 2025 Mar 17. PMID 40101437
- [Derived] Okuda R, Ogura T, Hisata S, Baba T, Kondoh Y, Suda T, Johkoh T, Iwasawa T, Tomioka H, Bando M, Azuma A, Inoue Y, Arai T, Nakamura Y, Miyamoto A, Miyazaki Y, Chiba H, Ishii H, Hamada N, Terasaki Y, Kuwahira I, Sato S, Kato S, Suzuki T, Sakamoto S, Nishioka Y, Hattori N, Hashimoto N, Morita S, Ichihara N, Miyata H, Hagiwara K, Nukiwa T, Kobayashi K. Design and rationale of the Japanese Idiopathic Interstitial Pneumonias (JIPS) Registry. Respir Investig. 2023 Jan;61(1):95-102. doi: 10.1016/j.resinv.2022.08.009. Epub 2022 Nov 15. PMID 36580379